CLINICAL TRIAL: NCT01887340
Title: Therapeutic Strategy Guided by PET-TDM for Patients With Grade I or Metastatic Seminoma
Brief Title: Therapeutic Strategy Guided by PET-TDM for Patients With Seminoma
Acronym: SEMITEP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2012-A01615-38; 2012/1884 (Other: CSET number)
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Seminoma
MeSH Terms: conditions — Seminoma | interventions — Carboplatin; Etoposide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): * PET-TDM
  * carboplatine: Dose (mg) = AUC x (GFR + 25)
    * GFR : glomérulaire filtration (ml/min)
    * AUC : area under curve (mg/ml x min)
  Interventions: Drug: Carboplatin
- Cohort 2 (Experimental): * PET-TDM
  * ETOPOSIDE (100 mg/m2 D1 to D5) and CISPLATINE (20 mg/m2 de D1 to D5)
  * carboplatine: Dose (mg) = AUC x (GFR + 25)
    * GFR : glomérulaire filtration (ml/min)
    * AUC : area under curve (mg/ml x min)
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Cisplatin

INTERVENTIONS:
Drug: Carboplatin — - carboplatine: Dose (mg) = AUC x (GFR + 25)
  * GFR : glomérulaire filtration (ml/min)
  * AUC : area under curve (mg/ml x min)
Drug: Etoposide — 100 mg/m2 D1 to D5
  Arms: Cohort 2
Drug: Cisplatin — 20 mg/m2 de D1 to D5
  Arms: Cohort 2

SUMMARY:
The purpose of the study is to evaluate the ration of patients getting an lighten therapeutic strategy after 18F-fluoro-désoxyglucose positron emission tomography (PET-TDM) in grade I (cohort 1) or metastatic (cohort 2) seminoma

ELIGIBILITY:
Inclusion Criteria shared:

* Histologically proved seminoma after orchiectomy
* Primary testicular or retroperitoneal
* Normal alpha-fetoprotein before and after orchiectomy
* No prior treatment with radiotherapy or chemotherapy
* Age >= 18 years
* ECOG 0 to 2
* PNN >= 1500, platelets >= 100 000, bilirubin <= the upper limit nromale
* ASAT (SGOT) and ALAT (SGPT) <= 1,5 x the upper limit nromale
* Serum creatinine <140 µmol / L (or clearance> 60 mL / min)
* Information and signed informed consent before inclusion in the study
* Patient affiliated to a social security

Specific inclusion criteria for cohort 1:

* grade I

Specific inclusion criteria for cohort 2:

* grade IIB (retroperitoneal adenopathy diameter between 2 cm and 5 cm, regardless of the LDH)
* grade IIC (retroperitoneal adenopathy diameter higher than 5 cm, regardless of the LDH)
* grade III of good prognosis (supradiaphragmatic reach with ganglionic metastasis and LDH < 2 times normal limit and/or supradiaphragmatic reach with pulmonary metastasis and LDH < 2 times normal limit) either at initial diagnosis or relapse of a grade I seminoma)
* PET-TDM positive (pathological fixation on metastatic lesions)

Exclusion Criteria shared:

* Patient infected by HIV, Hepatitis B or C
* History, within 5 years, of cancer other than seminoma, except for treated skin cancer (Basal Cell) .
* visceral metastasis
* cerebral metastasis
* Any physical or mental condition incompatible with the treatment (to the investigator discretion)
* Uncontrolled or severe cardiovascular pathology
* Uncontrolled or severe hepatic pathology
* Persons deprived of liberty or under guardianship
* Unable to undergo medical monitoring due to geographical, social or psychological reasons

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of patients without pathological fixation | Assessed at the time of inclusion or after 2 cycles of chemotherapy, up to 21 days
  Rate of patients without pathological fixation at the time of the inclusion PET-TDM (cohort 1) or at the time of the PET-TDM following two cycles of chemotherapy (Etoposiede+Cisplatine) (cohort 2) and getting a lighten protocol

SECONDARY OUTCOMES:
Rate of patients without pathological fixation | Assessed at the time of inclusion or after 2 cycles of chemotherapy, up to 21 days
  Rate of patients without pathological fixation at the time of the inclusion PET-TDM (cohort 1) or at the time of the PET-TDM following two cycles of chemotherapy (Etoposiede+Cisplatine) (cohort 2)
Progression Free Survival (PFS) | Assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yohann LORIOT, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France

REFERENCES:
- [Derived] Loriot Y, Texier M, Culine S, Flechon A, Thiery-Vuillemin A, Gravis G, Geoffrois L, Chevreau C, Gross-Goupil M, Barthelemy P, Bompas E, Mahammedi H, Laguerre B, Lacourtoisie SA, Helissey C, Ladoire S, Abraham C, Massard C, Grimaldi S, Fizazi K. The GETUG SEMITEP Trial: De-escalating Chemotherapy in Good-prognosis Seminoma Based on Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography. Eur Urol. 2022 Aug;82(2):172-179. doi: 10.1016/j.eururo.2022.04.031. Epub 2022 May 20. PMID 35599187